CLINICAL TRIAL: NCT04744792
Title: Quality of Life After Colorectal Surgery: A Prospective Study of Patients Compared With Their Spouses
Brief Title: QoL of Colorectal Cancer Patients and Spouses
Status: Completed | Type: Observational
Sponsor: Cihangir Akyol (Other)
Responsible Party: Sponsor-Investigator, Cihangir Akyol, Associate Proffessor, Ankara University
Organization: Ankara University (Other)
Other Study IDs: U1111-1264-6381
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Quality of Life; Stoma Ileostomy; Stoma Colostomy; Rectum Cancer; Sigmoid Cancer
Keywords: Quality of Life, SF - 36, Rectal cancer, spouse
MeSH Terms: conditions — Rectal Neoplasms; Sigmoid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: All the patients who underwent anterior resection, low anterior resection and abdominoperineal resection between march 2006 and novenmer 2010
  Interventions: Other: Short Form - 36; Other: WHODAS-II
- Spouses: Spouses of the patients who underwent anterior resection, low anterior resection and abdominoperineal resection between march 2006 and novenmer 2010
  Interventions: Other: Short Form - 36; Other: WHODAS-II

INTERVENTIONS:
Other: Short Form - 36 — Medical outcomes: 36-item short form health survey (SF-36)
  The SF-36 was used as a measure of health-related QoL because it is an internationally recognized global measure. It comprises 36 items that measure perceived health on eight scales (i.e., physical functioning, physical role, bodily pain, general health, vitality, social functioning, emotional role, and mental health) with higher scores (range 0-100) reflecting better perceived health. Additionally, two summary scores can be obtained: the physical component summary score (PCS) and the mental component summary score (MCS).
  In addition, this tool has been validated in Turkish patients
Other: WHODAS-II — The World Health Organization disability assessment schedule II (WHODAS-II)
  The WHODAS-II is an instrument developed by the World Health Organization to assess behavioral limitations and restrictions regarding participation in specific activity domains experienced by an individual independent of their medical diagnosis. The conceptual frame of reference of this instrument is the International Classification of Functioning, Disability, and Health (ICF). Specifically, the instrument is a 36-item, generic, multidimensional questionnaire designed to evaluate the functioning of the individual in six activity domains (i.e., understanding and communicating, getting around, self-care, getting along with people, life activities, and participation in society). This questionnaire has been validated in Turkish patients.

SUMMARY:
The aim of the present prospective, comparative study was to compare the quality of life (QoL) of patients after colorectal surgery to the QoL of their spouses. The study included patients who underwent curative surgery for colorectal carcinoma (n = 100; abdominoperineal excision [n = 33], low anterior resection [n = 33], left hemicolectomy [n = 34]) and their spouses (n = 100). The patients and spouses completed the Medical Outcome Study 36-item Short Form Survey (SF-36) and the World Health Organization Disability Assessment Schedule II (WHODAS-II) preoperatively and at postoperative months 15 to 18. The QoL of patients and that of their spouses changed following surgery for colorectal cancer.

These changes were more significant among male patients' spouses.

DETAILED DESCRIPTION:
There is no doubt that radical colorectal surgery improves the oncological outcomes of patients with cancer. However, the literature has clearly documented that social, physical, sexual, and psychological aspects of life, as well as religious worship, are severely impaired after this treatment. A significant portion of patients suffer from alterations in their quality of life (QoL), particularly after surgery on distal rectal tumors. Patients who require a stoma or who have low anterior resection syndrome may face difficulty adapting to their new anatomy, managing the stoma, defecating, and continuing normal activities in their sociocultural environment. Patients pay an immense price following both sphincter-saving and sphincter-sacrificing surgery. Moreover, these psychological and social difficulties, as well as sexual dysfunction, may affect patients' relationships with their spouses, who are generally the primary informal caregivers for patients with cancer. In addition to caring for their sick partners, the spouses also have to deal with their own anxiety, fatigue, and depression.The aim of the present prospective, comparative study was to compare the quality of life (QoL) of patients after colorectal surgery to the QoL of their spouses.

Groups

Patients and their spouses were grouped by the type of surgery they received:

abdominoperineal resection (APR), sphincter-saving resection with an anastomosis within 6 cm of the anal verge on rigid sigmoidoscopy (LAR), or anterior resection with anastomosis at or above 7 cm, including sigmoid colectomy (AR).

The study included patients who underwent curative surgery for colorectal carcinoma (n = 100; abdominoperineal excision [n = 33], low anterior resection [n = 33], left hemicolectomy [n = 34]) and their spouses (n = 100). The patients and spouses completed the Medical Outcome Study 36-item Short Form Survey (SF-36) and the World Health Organization Disability Assessment Schedule II (WHODAS-II) preoperatively and at postoperative months 15 to 18.

Counseling Surgical details, possible complications, and temporary or permanent stoma formation were explained preoperatively by the surgeon, and ostomy education was given by the stomatherapist. Religious education and counseling were also performed. Patients had direct access to doctors, the stomatherapist, appliance suppliers, and a religious leader (Imam) at the hospital during the study period.

Interviews Patients and spouses were interviewed at the Department of Surgery of Ibni Sina Hospital.

The coauthors of the study were trained to administer the questionnaires in a standard fashion and practiced by using the questionnaires on healthy volunteers before the study began.

Patients and spouses were interviewed in a private room by a person of the same gender. The same interviewer was used in the preoperative and postoperative period for each patient and spouse, but the interviewer was not blinded to the type of surgery that the patient had undergone. Patients were first asked to complete a demographic questionnaire designed to determine their age, gender, marital status, educational level, income level, and preoperative employment. The SF-36, WHODAS-II, and Ankara University Life Standards Questionnaire were administered together and consisted of a total of 92 items, which took approximately 35 to 45 minutes to complete. Both patients and spouses completed the SF-36, WHODAS-II, and Ankara University Life Standards Questionnaire preoperatively and at postoperative months 15 to 18.

ELIGIBILITY:
Inclusion Criteria:

1. curative surgery for colorectal adenocarcinoma
2. living with a spouse
3. aged over 18 years
4. Muslim faith.

Exclusion Criteria:

1) Other primary malignant tumors 4) Additional complicating or disabling disease that necessitated nursing assistance (e.g., mental illness) 5) Chemo-radiotherapy within 8 weeks prior to the interview 6) Admittance to a hospital except for stoma closure during the study period (no interview during stoma closure) 7) Major morbidity (e.g., anastomotic leakage, abdominal sepsis, stoma-related problems, and intensive care unit transfer) 8) Evidence of disease recurrence or metastasis, which was determined at the time of follow-up interviews

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had a spouse, aged 18 or over, and underwent abdominoperineal excision, low anterior resection, anterior resection between march 2006 and november 2010 in Ankara University Department of general surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2006-03-01 (Actual); Primary Completion 2010-11-01 (Actual); Study Completion 2010-11-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life of patients and spouses | In the preoperative period
  Medical outcomes: 36-item short form health survey (SF-36)
  The SF-36 was used as a measure of health-related QoL because it is an internationally recognized global measure. It comprises 36 items that measure perceived health on eight scales (i.e., physical functioning, physical role, bodily pain, general health, vitality, social functioning, emotional role, and mental health) with higher scores (range 0-100) reflecting better perceived health. Additionally, two summary scores can be obtained: the physical component summary score (PCS) and the mental component summary score (MCS).
Quality of Life of patients and spouses | postoperative 15th month
  Medical outcomes: 36-item short form health survey (SF-36)
  The SF-36 was used as a measure of health-related QoL because it is an internationally recognized global measure. It comprises 36 items that measure perceived health on eight scales (i.e., physical functioning, physical role, bodily pain, general health, vitality, social functioning, emotional role, and mental health) with higher scores (range 0-100) reflecting better perceived health. Additionally, two summary scores can be obtained: the physical component summary score (PCS) and the mental component summary score (MCS).
Disability of patients and spouses | In the preoperative period
  The World Health Organization disability assessment schedule II (WHODAS-II)
  The WHODAS-II is an instrument developed by the World Health Organization to assess behavioral limitations and restrictions regarding participation in specific activity domains experienced by an individual independent of their medical diagnosis. The conceptual frame of reference of this instrument is the International Classification of Functioning, Disability, and Health (ICF). Specifically, the instrument is a 36-item, generic, multidimensional questionnaire designed to evaluate the functioning of the individual in six activity domains (i.e., understanding and communicating, getting around, self-care, getting along with people, life activities, and participation in society).
Disability of patients and spouses | postoperative 15th month
  The World Health Organization disability assessment schedule II (WHODAS-II)
  The WHODAS-II is an instrument developed by the World Health Organization to assess behavioral limitations and restrictions regarding participation in specific activity domains experienced by an individual independent of their medical diagnosis. The conceptual frame of reference of this instrument is the International Classification of Functioning, Disability, and Health (ICF). Specifically, the instrument is a 36-item, generic, multidimensional questionnaire designed to evaluate the functioning of the individual in six activity domains (i.e., understanding and communicating, getting around, self-care, getting along with people, life activities, and participation in society).

CONTACTS AND LOCATIONS:
Overall Officials: cihangir Akyol, Study Director — Ankara University School of Medicine Departmernt of General Surgery